CLINICAL TRIAL: NCT03107533
Title: Scoliosis Shared Decision Making
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, A. Noelle Larson, MD, Associate Professor of Orthopedics, Mayo Clinic
Other Study IDs: 17-002245
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Video recording of clinical visit: Investigators will enroll patients from the Department of Orthopedic Surgery for enrollment. The shared decision group will provide staff for data analysis.
  Interventions: Other: Video recording of clinical visit

INTERVENTIONS:
Other: Video recording of clinical visit — For patients and parents that are considering scoliosis surgery, a video recording of the encounter will be obtained during their routine clinical visit to discuss surgery/options.

SUMMARY:
Analysis of video encounters between providers, patients, and families will be used to develop a shared decision making tool for patients deciding between surgery and observation for scoliosis treatment.

DETAILED DESCRIPTION:
For patients and parents who are considering scoliosis surgery, a video recording of the encounter will be obtained during their routine clinical visit to discuss surgery/options. This video will then be sent to the shared decision making group at Mayo Clinic, Rochester, Minnesota to run analysis of the data (Shared Decision Making National Resource Center, Knowledge and Evaluation Research Unit, Mayo Clinic). Investigators will follow the patient's electronic medical records for 2 years after their decision of treatment option. No outcome forms will be specifically collected as part of the study, as outcomes forms are currently being collected clinically on all scoliosis patients.

Based off of the initial video recordings, the first visual prototype of the shared decision making tool for scoliosis has been developed. This prototype of the shared decision making tool will be now be used to help test it's efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis curve >40 degrees, < 65 degrees
* Risser score > 2
* Age > 13 years

Exclusion Criteria:

* Risser score of 0 or 1
* Non-ambulatory scoliosis patients
* Ages 12 year and under

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who understand disease treatment as determined by analysis of video recording | Baseline
  Video will be recorded then be sent to the shared decision making group at Mayo Clinic, Rochester, Minnesota to run analysis of the data (Shared Decision Making National Resource Center, Knowledge and Evaluation Research Unit, Mayo Clinic).

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Larson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials